CLINICAL TRIAL: NCT05700929
Title: Evaluation of a Patient-centered Communication Skills Training for Nursing Professionals in Germany: A Randomized Controlled Trail
Brief Title: Evaluation of a Communication Skills Training for Nurses
Acronym: KOMPAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Isabelle Scholl, Prof.Dr., Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1047/136
Record Dates: First submitted 2022-11-16; First posted 2023-01-26 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Communication
Keywords: Nursing; Communication skills; Communication skills training; Patient-centered; Train-the-trainer; Health Services Research; Implementation Research; Hybrid type 1 effectiveness-implementation trial; Randomized controlled trial; Mixed Methods; Self-Efficacy
MeSH Terms: conditions — Communication | interventions — Nurses

STUDY DESIGN:
Intervention Model Description: This study is a hybrid type 1 effectiveness-implementation trial, conducted as a two-armed randomized controlled trial including a comprehensive process evaluation for future implementation. After baseline assessment, participants will be randomized to the intervention group or the waitlist-control group. Randomization will be performed using stratified permuted block randomization. The waitlist-control group are offered to participate in the communication skills training after data collection has been finished.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Communication skills training (Experimental): The intervention is a one-day face-to-face training to foster patient-centered communication skills of nursing professionals at the University Medical Center Hamburg-Eppendorf, Germany. The training is developed based on results of a previously conducted needs assessment with nurses, medical assistants and nursing service managers as well as literature research and will be rolled out after baseline assessment and randomization.
  Interventions: Behavioral: Communication skills training for nurses
- Waitlist-control group (No Intervention): Participants of the waitlist-control group receive no specific study related intervention. Participants of this group will be offered a communication skills training after complete data collection of all participants of the RCT has been finished.

INTERVENTIONS:
Behavioral: Communication skills training for nurses — Aim of the developed training will be to foster patient-centered communication skills of nursing professionals in Germany. The training consists of four modules in which participating nurses will get information regarding patient-centeredness and general communication techniques. Participants will also learn how to response to patients in escalating situations and how to communicate with seriously ill or dying patients. The underlying framework for the training is the Calgary-Cambridge Guide, a well-known model for structuring conversation with patients. Different didactic techniques (i.e. roll-play, video sequences, group discussion) will be applied. The training will be provided in small groups of 10-14 participants each. Two facilitators will give the training, one of them being a nursing professional trained according to the train-the-trainer approach, the other being a member of the research group, who was involved in the development of the training.
  Arms: Communication skills training

SUMMARY:
The KOMPAT study aims to evaluate the effectiveness and feasibility of a needs-based communication skills training for nursing professionals in Germany and to derive recommendations for future long-term implementation. Therefore, a training program to foster communication skills of nursing professionals has been developed based on a previously conducted needs assessment and literature research. To evaluate the training a randomized controlled trail with a waitlist-control group will be conducted. It is aimed to include 180 nurses within the study, of which 90 nurse will be randomized in a stratified manner to the intervention group and 90 nurses will be randomized to the waitlist-control group. Outcomes will be assessed at baseline, post -training and 4-weeks follow-up. It is hypothesized that self-efficacy in communication with patients and further outcomes will be significantly higher among participants in the intervention group compared to participants of the waitlist-control group during post-training assessment and follow-up. The evaluation will be accompanied by a process evaluation. The training will be facilitated by a member of the research team and a nursing professional by applying the train-the-trainer approach. The KOMPAT study will be conducted at the University Medical Center Hamburg-Eppendorf.

ELIGIBILITY:
Inclusion Criteria:

* Nurses working at the participating departments of the University Medical Center Hamburg-Eppendorf
* Main part of daily work includes communication with patients
* Age ≥ 18 years
* Completed educational program as a nurse
* German-speaking

Exclusion Criteria:

* Little or no contact with patients in daily work, e.g. an operating room nurse or within the bed management

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Self-efficacy regarding communication with patients | Change from baseline (t0) at immediately after the training (t1) (with t1 being the primary endpoint) and at four weeks after the training (t2) for the intervention and waitlist-control group.
  Description: Self-efficacy of nurses in the context of communication with their patients will be measured by the German version of the 12-item Self-Efficacy Scale (SE-12-G). Items on this one-dimensional scale can be answered on a scale from 1 ("very uncertain") to 10 ("very certain") with an additional option to rate items as "not relevant".

SECONDARY OUTCOMES:
Rating of the training | immediately after the training (t1) for the intervention group
  Rating of the training by participating nurses according to the trainings' content, used materials and didactic, measured by a short self-developed scale adapted from previous studies on the evaluation of communication skills trainings at the University Medical Center Hamburg-Eppendorf.
Subjective knowledge about patient-centered communication | Change from baseline (t0) at immediately after the training (t1) and at four weeks after the training (t2) for the intervention and waitlist-control group
  Assessment of nurses' subjective knowledge regarding patient-centered communication topics, which will be conveyed in the trainings, measured by a short self-developed scale adapted from a previous study of the research team and adapted to the content of the communication skills training.
Objective knowledge about patient-centered communication | Change from baseline (t0) at immediately after the training (t1) and at four weeks after the training (t2) for the intervention and waitlist-control group
  Assessment of nurses' objective knowledge regarding patient-centered communication topics, which will be conveyed in the trainings, measured by several multiple choice questions developed according to the content of the communication skills training.
Attitudes towards medical communication | Change from baseline (t0) at four weeks after the training (t2) for the intervention and waitlist-control group
  Assessment of nurses' attitudes towards medical communication measured via the German version of the 12-item Attitudes towards medical communication scale (ATMC-G).
Communication skills of nurses from external observers' perspective after participation in a SPA | four weeks after the training (t2) for the intervention and waitlist-control group
  Objective rating of nurses' communication skills measured via Standardized Patient Assessments (SPAs). Content of SPAs were developed according to the content of the communication skills training. Ratings will be conducted by one trained member of the research team who has not previously trained the participants. Additionally, the level of anxiety associated with performing in a SPA will be assessed via the subscale 'cognitive anxiety' and the subscale 'physiological anxiety' of the Performance Text Anxiety questionnaire (PTA).
Communication skills of nurses from simulation patients' perspective after participation in a SPA | four weeks after the training (t2) for the intervention and waitlist-control group
  After SPAs, simulation patients will assess their perceived patient-centeredness during the SPA situation with the participating nurse using items of the dimensions 'communication' and 'patient-centerdness' of the German measure Experienced Patient-Centeredness Questionnaire (EPAT).
Self-assessed communication skills from participants' perspective after participation in a SPA | four weeks after the training (t2) for the intervention and waitlist-control group
  After SPAs, the participating nurses will self-assess their perceived communication skills via several items of the long version of the German measure Experienced Patient-Centeredness Questionnaire (EPAT), adapted for healthcare professionals.
Professional fulfillment | Change from baseline (t0) at immediately after the training (t1) and at four weeks after the training (t2) for the intervention and waitlist-control group
  Job-related psychological burden of participating nurses including professional fulfillment, work exhaustion, interpersonal disengagement and overall burnout, measured via the German version of the 16-item Professional Fulfillment Index (PFI-G).
Depression and anxiety | Change from baseline (t0) at immediately after the training (t1) and at four weeks after the training (t2) for the intervention and waitlist-control group
  Depression and anxiety will be measured using the German version of the 4-item measure Patient Health Questionnaire 4 (PHQ-4).
Subjective working capacities | Change from baseline (t0) at immediately after the training (t1) and at four weeks after the training (t2) for the intervention and waitlist-control group
  Subjective working capacities of participating nurses, measured via three items covering the first two dimensions of the German version of the Work Ability Index (WAI).
Experienced patient-centeredness (Covariate) | Change from baseline (t0) at four weeks after the training (t2) for the intervention and waitlist-control group
  Experienced person-centered climate on the wards, assessed by healthcare professionals working on the wards, measured via an adapted version of the German 16-item measure Experienced Patient-Centeredness Questionnaire (EPAT).
Impact of contamination (Covariate) | for the intervention group at baseline (t0) only; for the waitlist-control group at baseline (t0), immediately after the training (t1) and four weeks after the training (t2)
  The measure the extent to which participants have received information about the training content prior to participation or for the waitlist-control group during all measurement points from participants, who participated already in the training, a self-developed item on the impact of contamination will be used.

OTHER OUTCOMES:
Process evaluation | through study completion and until approximately June 2025
  Assessment of the implementation process applying the Consolidated Framework for Implementation Research (CFIR) to describe fidelity and reach by documenting the implementation of the study, taking field notes by taking field notes while conducting the study as well as acceptability and appropriateness of the intervention by conducting semi-structured interviews with relevant stakeholders including non-participants of the study.
Demographic items | baseline (t0) for the intervention and waitlist-control group
  Assessment of basic demographic information including age, sex, function, work experience, previous experience with communication skills trainings .

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lindig A, Mielke K, Frerichs W, Collen K, Kriston L, Harter M, Scholl I. Evaluation of a patient-centered communication skills training for nurses (KOMPAT): study protocol of a randomized controlled trial. BMC Nurs. 2024 Jan 2;23(1):2. doi: 10.1186/s12912-023-01660-8. PMID 38163904
- See also: Related Info — http://www.uke.de/kliniken-institute/institute/institut-und-poliklinik-für-medizinische-psychologie/forschung/arbeitsgruppen/kompat-projekt.html